CLINICAL TRIAL: NCT04329715
Title: Expedited Versus Restrictive: Limitations on Activity Following Surgical Treatment of Prolapse
Acronym: EVeRLAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00104389
Record Dates: First submitted 2020-03-30; First posted 2020-04-01 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Intervention Model Description: Randomized controlled non-inferiority trial
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Surgical treatment teams and outcome assessors will be blinded to patient's treatment arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Expedited instructions (Experimental)
  Interventions: Behavioral: Expedited postoperative activity instructions
- Restricted instructions (Active Comparator)
  Interventions: Behavioral: Standard postoperative activity restructions

INTERVENTIONS:
Behavioral: Expedited postoperative activity instructions — Ad lib postoperative activity and return to work recommendations
  Arms: Expedited instructions
Behavioral: Standard postoperative activity restructions — Standard conservative postoperative activity and return to work recommendations
  Arms: Restricted instructions

SUMMARY:
The objective of the EVeRLAST study is to determine whether expedited resumption of postoperative activity levels is non-inferior to standard activity restrictions with respect to short-term anatomic prolapse outcomes. We hypothesize that immediate resumption of physical activities as tolerated will result in noninferior surgical outcomes following prolapse surgery when compared to standard postoperative activity restrictions.

Participants will be enrolled and randomized at their preoperative clinic visit to one of two treatment arms:

Arm 1: Standard instructions (no heavy lifting over 10lbs for 6 weeks; return to work at 4 weeks for sedentary work and 6 weeks for manual labor) Arm 2: Liberal instructions (no restrictions; resume activities and work as soon as able)

We will also collect subjective and objective measures of pre- and postoperative physical activity, through the use of patient-reported physical activity assessments and wrist-worn accelerometers. Accelerometer data will be collected at the preoperative, 2-week-postoperative, and 6-week-postoperative time points. Accelerometer data will also be used to calculate time to resumption of normal activities, defined as time at which a patient resumes greater than 90% of her baseline preoperative level of physical activity. We will additionally be collecting data on relevant patient-reported outcomes of pelvic floor symptom severity, health-related quality of life measures, postoperative pain, time to return to work (where relevant), and patient global impression of improvement. Postoperative anatomic assessments will be performed at 6 weeks and 3 months postoperatively by blinded study personnel

DETAILED DESCRIPTION:
Specific aim 1: Determine if liberal (ad lib) resumption of postoperative activity levels is non-inferior to standard restrictions with regards to short-term anatomic and symptomatic outcome, as measured by maximum pelvic organ prolapse support loss ('SLmax') and the Pelvic Organ Prolapse Distress Inventory (POPDI) at 3 months. (Co-primary outcome)

Specific aim 2: Compare postoperative "Recovery Time" and physical function between women instructed to resume their activity levels ad lib versus women instructed to restrict activity levels. "Recovery Time," defined as the postoperative day at which the patient resumes 90% of her baseline activity levels will be objectively measured using the Actigraph accelerometer.8 ,9 Physical function will be measured with the 6-minute walk, chair stand tests, and through patient-reported outcome measures. (exploratory outcome)

Specific aim 3: Compare timing of return-to-work and health-related QOL in women instructed to resume activity levels and return to work ad lib versus restrict their activity levels (exploratory outcome)

Eligible participants will first be briefly explained regarding the research study. If interested, will then complete the informed consent process. She will first be asked to complete the International Physical Activity Short Form to confirm study eligibility. For study eligibility, participants must at least report a baseline of 725 MET-minutes per week of physical activity according to the IPAQ-SF, which is consistent with the lowest quartile of activity among elderly women. If she reports greater than 725 MET-minutes per week of physical activity, she will undergo the remainder of baseline assessments. If she reports less than 725 MET-minutes per week of physical activity, she will be explained that she does not meet the activity level criteria for completion of the study at this time. She will then be asked to complete a series of baseline questionnaires (demographics, past medical history, POPDI, AAS, PROMIS, PFDI, PFIQ). She will also undergo a baseline POPQ exam and tests of physical function, including the 6-minute walk test and chair stand test.

A sealed envelope will then be opened by the research coordinator (or study investigator) in front of the patient indicating the patient's study allocation. The packet will also include an accelerometer which the patient will be instructed to wear for a 7-day period preoperatively. However, to ensure that participants are not given an accelerometer too far in advance from her surgery (as at times surgery may be scheduled remotely from the initial decision to proceed with surgery which would potentially result in too many accelerometers being out of circulation), the envelope containing study allocation and accelerometers may alternatively be provided at the preoperative "Surgical Workup" visit once the surgery is scheduled and at a date no greater than 3 weeks from the planned surgery. If a participant will be undergoing surgery at an interval greater than 1 week from the initial receipt of the accelerometer, she will only be required to wear the accelerometer for 1 week prior to the surgery. Patients will be given an opportunity to ask any questions regarding postoperative activity instructions to research personnel or nurses at the time of study enrollment and at any point prior to her surgery. Patients will be notified, prior to providing consent, that her primary surgeon will remain blinded as to her treatment allocation until completion of her study participation.

Any questions related to surgical recovery which arise preoperatively will be addressed by nurses and research personnel not involved in the patient's intraoperative decision-making. Postoperatively, fellow and attending surgeons will only be unblinded if necessary to address any acute postoperative issues. Patients will also be provided with a duplicate set of postoperative set of activity instructions on the day of her surgery upon discharge which will be entered in the patient's electronic chart by study personnel on the day of her surgery as a modification to the standard postoperative discharge instructions.

The patient will wear the activity tracker for 6 weeks postoperatively. At the 1-week postoperative time point, patient reminder phone calls will be made to remind the patient to wear and charge the activity tracker (whose battery life is 25 days). She will also be asked to provide a count of the number of narcotic pills she has left remaining at this time. She will follow-up for a routine postoperative visit with her primary surgeon at which point a routine 6-week postoperative POPQ will be performed. Accelerometers will be returned at this visit.

She will then follow up for a separate research visit at 3 months postoperatively. At this time, the patient will complete all follow-up activity, symptom, and HRQOL questionnaires including the: Activities Assessment Scale, Pelvic Floor Distress Inventory, Pelvic Floor Impact Questionnaire, and the PROMIS short form subscales of physical function, anxiety, depression, fatigue, satisfaction with social role, and pain interference. A six-minute walk and chair stand test will be administered by trained research personnel in the clinic. She will additionally be inquired regarding timing of return to work. A POPQ will also be performed at this time by a blinded provider NOT involved in the patient's index surgery.

ELIGIBILITY:
Inclusion Criteria:

* Stage II-IV pelvic organ prolapse
* Bothersome bulge symptoms
* At least 725 MET-minutes/week on International Physical Activity Questionnaire Short Form
* English-speaking
* Undergoing treatment of prolapse
* Surgery occurring at least 7 days from date of randomization (to allow for collection of at least 7 days of preoperative accelerometer data)
* Able and willing to follow up at 3 months for in-office exam

Exclusion Criteria:

* Enrollment in another research study of pelvic organ prolapse
* Concomitant non-urogynecologic surgery
* Planned further surgery in the next 3 months or anticipated treatment which would result in prolonged inactivity (such as a cancer diagnosis) 3 months postoperatively

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Maximum support loss "SLMax" | 3 months
  Most distal point of pelvic organ support (in centimeters) based on Pelvic Organ Prolapse Quantification system
Prolapse symptoms | 3 months
  Pelvic Organ Prolapse Distress Inventory (POPDI) at 3 months

SECONDARY OUTCOMES:
Recovery time | 6 weeks
  Time to resumption of >90% of baseline activity, measured with ActiGraph accelerometer worn pre- and 6 weeks postoperatively
Health related quality of life (HRQOL) | 3 months
  HRQOL as measured by the PROMIS short form subscales of physical function, anxiety, depression, fatigue, satisfaction with social role, and pain interference
Physical function | 3 months
  Functional aerobic capacity as measured by the 6 Minute Walk Test
Physical function | 3 months
  Functional strength as measured by the Chair Stand Test
Time to return to work | 3 months
  Postoperative day at which patient returned to work
Postoperative opioid requirement | 2 weeks
  Opioid pill count
Pelvic floor symptom severity | 3 months
  Measured by the Pelvic Floor Distress Inventory-20
Pelvic floor symptom severity | 3 months
  Measured by the Pelvic Floor Impact Questionnaire-7
Functional activity | 3 months
  As measured by the Activities Assessment Scale
Patient satisfaction | 3 months
  As measured by Patient Global Impression of Improvement
Postoperative morbidity | 3 months
  Postoperative morbidity following surgery

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Barber, MD, MHS, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brubaker L, Barber MD, Nygaard I, Nager CW, Varner E, Schaffer J, Visco A, Meikle S, Spino C; Pelvic Floor Disorders Network. Quantification of vaginal support: are continuous summary scores better than POPQ stage? Am J Obstet Gynecol. 2010 Nov;203(5):512.e1-6. doi: 10.1016/j.ajog.2010.06.071. Epub 2010 Aug 21. PMID 20728072
- [Background] Tomioka K, Iwamoto J, Saeki K, Okamoto N. Reliability and validity of the International Physical Activity Questionnaire (IPAQ) in elderly adults: the Fujiwara-kyo Study. J Epidemiol. 2011;21(6):459-65. doi: 10.2188/jea.je20110003. Epub 2011 Sep 24. PMID 21946625
- [Derived] O'Shea M, Siddiqui NY, Truong T, Erkanli A, Barber MD. Standard Restrictions vs Expedited Activity After Pelvic Organ Prolapse Surgery: A Randomized Clinical Trial. JAMA Surg. 2023 Aug 1;158(8):797-805. doi: 10.1001/jamasurg.2023.1649. PMID 37256578